CLINICAL TRIAL: NCT07041645
Title: Bioavailability of Micronutrients With a Special Focus on Vitamin K - Study Part I: K-vitamin
Brief Title: Bioavailability of Different Vitamin K Vitamers Studied Using 13C-labelled Vitamin K Vitamers
Acronym: BioMicro
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Technical University of Denmark (Other)
Responsible Party: Principal Investigator, Susanne Bügel, Professor, Head of Section, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: BioMicro Protokol v1.2
Record Dates: First submitted 2025-06-19; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Bioavailability of Vitamin K
Keywords: Bioavailability; vitamin K; 13C-labelled vitamin K
MeSH Terms: interventions — Vitamin K

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 13C-phylloquinone (13C-PK) (Experimental): The participants will receive one dose of 13C-PK and the levels in blood, urine and feces will be analyzed
  Interventions: Dietary Supplement: Vitamin K
- 13C-menaquinone-4 (13C-MK-4) (Experimental): The participants will receive one dose of 13C-MK-4 and the levels in blood, urine and feces will be analyzed
  Interventions: Dietary Supplement: Vitamin K
- 13C-menaquinone-7 (13C-MK-7) (Experimental): The participants will receive one dose of 13C-MK-7 and the levels in blood, urine and feces will be analyzed
  Interventions: Dietary Supplement: Vitamin K
- 13C-menaquinone-9 (13C-MK-9) (Experimental): The participants will receive one dose of 13C-MK-9 and the levels in blood, urine and feces will be analyzed
  Interventions: Dietary Supplement: Vitamin K

INTERVENTIONS:
Dietary Supplement: Vitamin K — each participant will recive one dose of each of the four vitamin K vitamers but in different orders (4 different orders).

SUMMARY:
Objectives

The main objectives are:

Study part I: to investigate the bioavailability of vitamin K vitamers (PK, MK-4, MK-7 and MK-9) in humans using 13C-labelled compounds

Hypotheses Study part I: it is hypothesized that there is a difference between the bioavailability of the different vitamers, with MK-9 having the highest bioavailability followed by MK-7, and then PK, while MK-4 will have the lowest bioavailability.

Participants will:

Study part I: In the pilot study and study part I, participants will visit NEXS for a test period where a 6.5-hour test day will be carried out and followed up with two short visits on the 2 consecutive days. In the pilot study, there will be one test period with frequent blood sampling (before and after ingestion of a labelled vitamin K vitamer) and urine and faeces sampling. The minimum duration for each participant in the pilot study will be 2.5 weeks. After analyses of the bioavailability of the vitamin K vitamers in the pilot study, results will be used to determine the time points for biological sampling (mainly blood) in study part I. Study part I is a cross-over study with 4 test periods and washout periods in between. The minimum duration for each participant will be 6 weeks.

DETAILED DESCRIPTION:
Overall study design Pilot study (n= 2 completers): An acute postprandial randomised parallel study comparing the bioavailability of two forms of labelled vitamin K vitamers (13C-PK and 13C-MK-7) Study part I (n= 16 completers): An acute postprandial randomised cross-over study comparing the bioavailability of four forms of labelled vitamin K vitamers (13C-PK, 13C-MK-4, 13C-MK-7, and 13C-MK-9)

Detailed study design of pilot study and part I Prerequisites

Prior to the first test period (day 0) the participants will be asked to:

* 2 weeks before: supplement with 10 µg vitamin D3/day (recommended daily intake) and restrain from all other types of (vitamins and mineral) supplementation
* 1 week before: not consume sweet corns, beetroot and spinach
* 48 hours before: alcohol intake is prohibited
* 24 hours before: high-intensity physical activity is prohibited
* 12 hours before: except 0.5 L tap water, consumption of drinks and foods are not allowed After the first test day and during the remaining part of the study, the participants are asked to refrain from consumption of sweet corn, beetroot and spinach, continue supplementation with vitamin D. Before all days with blood sampling (3 first days in a test period), the above prerequisites related to alcohol intake, high-intensity physical activity and fasting are applicable.

Test periods A baseline description (e.g. anthropometry, blood pressure and fasting values) of the participants will be established prior to and on the first test day (Day 0).

In the pilot study, there will be one test period (Day 0-2) and in the study part I there will be four test periods (Day 0-2, 7-9, 14-15 and 21-23). Except for a few baseline outcomes only collected at Day 0, all test periods will follow the same overall design.

On the first day in a test period (e.g. Day 0), the participants will arrive fasting at NEXS, where a peripheral venous catheter (PVC) will be placed. The participants will rest for 10 minutes before the first blood sample will be taken in the fasting state ("0" minutes). The participants will hereafter have 15 minutes to ingest a breakfast meal containing a 13C-labelled vitamin K vitamer. Postprandial blood samples will hereafter be collected during a 5.5-hour period at the following time points after the breakfast was initiated: 15, 30, 45, 60, 90, 150, 210, 270 and 330 minutes. Furthermore, on the 2 consecutive days a fasting blood sample will be collected corresponding to 24 (±2) hours and 48 (±2) hours after the ingestion of the 13C-labelled vitamin K vitamer.

Results from the pilot study will be used to decide which biological sampling time points that are necessary in study part I where a maximum blood volume per test period will be 125 mL (for all 4 test periods the maximum blood volume will be 500 mL).

Wash out period Participants in the pilot study will have one washout period and participants in study part I will have 4 washout periods. During washout, the participants do not ingest the 13C-labelled vitamin K vitamer. In part I, the washout periods are minimum 6 days to ensure no carry over to the next administration period. Optimally, these washout periods will be planned at days: 1-6 (test period

1), 8-13 (test period 2), 15-20 (test period 3) and 22-27 (test period 4) and the participants will continue the collection of urine and faecal samples during the washout period. On day 7, participants in part I will repeat the test period (except the run-in period) and thus it continues until all 4 vitamin K vitamers have been tested.

In case of illness, vacations, holidays or practical project management reasons, the washout period can be extended. Extension of the washout period is not defined as a protocol deviation if all biological samples are collected on the consecutive days according to time points/definitions.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Between 18 and 65 years old (including both 18 and 65 year olds)
* Danish-speaking
* Willingness to consume/comply with consumption of study-related intervention products/diet
* Willing to take 10 µg vitamin D3/day and omit intake of all other (vitamins and mineral) supplements before and during the trial
* BMI ≤ 30.0 kg/m2

Exclusion Criteria:

* Daily smokers/users of all kinds of nicotine-containing products. Occasional smokers/user can be included if they are willing to refrain from all kinds of nicotine-containing products during the trial (from screening to end of trial)
* Blood donation <3 months prior to study-related blood sampling
* Intensive physical training (> 10 hours of strenuous physical activity per week)
* Participation in other clinical studies at the time of the study
* Pregnant, lactating or planning to become pregnant within the study period
* Habitual alcohol intake above current recommendation (> 10 alcoholic units/week)
* History of cancer within the past five (5) years except basal cell skin cancer and cervix
* Diagnosed with chronic inflammation disorders
* Diagnosed with gastrointestinal diseases
* Diagnosed with bone related diseases
* Diagnosed with psychiatric disorder including depression that requires medical treatment
* Medical treatment of diabetes
* Medical treatment of cardiovascular related disease
* Surgical change of the gastrointestinal tract (removal of appendix is allowed)
* Use of prescription medication that can affect their safety or impact on data
* Inability, physically or mental, to comply with the procedure required by the study protocol and evaluated by the principal investigator (PI), study manager or clinical responsible
* Medical treatment with anticoagulation medication (warfarin-like types)
* Allergy or intolerance related to intervention products

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
13C-labelled vitamin K vitamers in blood samples | from test day 1 until the end of the last washout period 5 weeks after test day 1.
  The area under the curve for the different 13C-labelled vitamin K vitamers will be compared from blood samples.
13C-labelled vitamin K vitamers in fecal samples | from test day 1 until the end of the last washout period 5 weeks after test day 1.
  The amount of 13C-labelled vitamin K vitamers in the feces will be analysed
13C-lebelled vitamin K vitamers in urine samples | from test day 1 until the end of the last washout period 5 weeks after test day 1.
  The amount of 13C-labelled vitamin K vitamers in the urine will be analysed

CONTACTS AND LOCATIONS:
Overall Officials: Susanne G Bügel, Professor, Principal Investigator — University of Copenhagen
Locations (1):
- University of Copenhagen, Frederiksberg C, Denmark

IPD SHARING:
Plan to Share IPD: No
We will report anonymized data for publications of the result.